CLINICAL TRIAL: NCT03669835
Title: The Sublimated Mare Milk Supplement In Patients With Hepatitis C
Brief Title: The Sublimated Mare Milk Supplement in Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Collaborators: Eurasia Invest Ltd. (Industry); Ministry of Education and Science, Republic of Kazakhstan (Other Government)
Responsible Party: Principal Investigator, Yermekbayeva Bakytgul, Principal Investigator, MD, PhD, Asfendiyarov Kazakh National Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KazNMU.MM.HC
Record Dates: First submitted 2018-09-06; First posted 2018-09-13 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Mare milk; Liver function
MeSH Terms: conditions — Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement and standard therapy. (Experimental): Participants will take a supplement of 1 sachet (20 mg) 3 times/day accompanied with the standard therapy for 1 month.
  Interventions: Dietary Supplement: Mare milk supplement; Drug: Standard therapy
- Standard therapy only. (Other): Patients would be given standard treatment for 1 month.
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Dietary Supplement: Mare milk supplement — Supplement consisting of sublimated mare's milk with single-dose 20 mg sachet. The supplement is dissolved in 36-27 degrees of Celsius water and taken 15-20 minutes before meal.
  Arms: Dietary supplement and standard therapy.
Drug: Standard therapy — For hepatitis virus C genotype 1: sofosbuvir 400 mg + lepidavir 90 mg for 12 weeks OR sofosbuvir 400 mg + daclatasvir 60 mg for 12 weeks; For hepatitis virus C genotypes 2 and 3: sofosbuvir 400 mg + daclatasvir 60 mg for 12 weeks.

SUMMARY:
This clinical trial studies the effect of sublimated mare milk supplement on patients with hepatitis C.

DETAILED DESCRIPTION:
Chronic viral hepatitis C is one of the medical, social and economic public health problems throughout the world. In majority of patients with chronic viral hepatitis C, dysbiotic changes are detected in the intestinal tract. Disturbances of microbial equilibrium are associated with the degree of inflammation, morphological changes in the liver, nature of the course and the stage of the disease.

These dysbiotic changes and and associated immune disorders can significantly aggravate the course of immune processes in the liver, converting hepatitis C infection to a chronic disease.

Mare milk is frequently reported for having therapeutic and dietary properties, which are initially associated with a specific chemical composition and certain physical properties of the product. It contains a total of about 40 biologically active components, the most important of them vitamins A, C, B1, B2, B6, B12, amino acids, enzymes and trace elements, there are low molecular weight peptides, lactalbumins and globulins.

The use of mare milk can contribute to the restoration of impaired functions of damaged organs and tissues, and play the role of an auxiliary pathogenetic therapy, primarily in certain chronic diseases of the digestive system, including chronic viral hepatitis C. Mare milk can also be used as a powder supplement through sublimation process.

In this trial, the effect of this supplement consisting of sublimated mare milk on hepatitis C patients will be evaluated. There will be two parallel groups: Interventional (sublimated mare milk supplement with standard treatment) and Standard treatment group. Differences in laboratory characteristics will be quantitively analyzed between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with verified diagnosis of hepatitis C
* Aged 18 to 65 years
* Normal intestinal microbiota composition (anaerobes-95%, aerobes-5%)
* Normal level of immune system markers in blood (Immunoglobulin M and Immunoglobulin G)
* Decreased levels of phosphatidylethanolamine, phosphatidylserine, phosphatidylcholine, sphingomyelin
* Elevated lysophosphatidylcholine
* Willingness to consent to participate in the study
* Consent to adhere to treatment

Exclusion Criteria:

* Drug and/or alcohol dependence
* Allergy to dairy products
* People with mental disabilities and/or life-threatening conditions
* Pregnancy and/or lactation
* Lactose intolerance
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in liver function. | Baseline, 2 weeks, 4 weeks, 8 weeks
  Change in liver function will be assessed from biochemical blood results of alanine transaminase and aspartate transaminase.
Change in urine test. | Baseline, 2 weeks, 4 weeks, 8 weeks
  Proportion of patients with deviations from normal range of urine test.

SECONDARY OUTCOMES:
Changes in gut microbiota composition. | Baseline, 2 weeks, 4 weeks, 8 weeks
  Proportions of aerobic and anaerobic bacteria will be assessed from stool samples using MiSeq Sequencing System.
Intestinal immune status changes. | Baseline, 2 weeks, 4 weeks, 8 weeks
  Level of immune status markers (Immunoglobulin G, Immunoglobulin M) will be detected from blood samples.
Changes in phospholipids spectrum of lymphocyte membranes. | Baseline, 2 weeks, 4 weeks, 8 weeks
  Detection of changes in phospholipids spectrum of lymphocyte membranes (phosphatidylethanolamine, phosphatidylserine, phosphatidylcholine, sphingomyelin, lysophosphatidylcholine) will be performed using the thin-layer chromatography method.
Changes in degree of liver fibrosis. | Baseline, 2 weeks, 4 weeks, 8 weeks
  Liver fibrosis will be evaluated using transient elastography method.

CONTACTS AND LOCATIONS:
Locations (1):
- Asfendiyarov Kazakh National Medical University, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yershova IB. Features of intestinal micro-biocenosis in viral hepatitis and possibilities of its correction. Actual Infectology 2(3): 7-11, 2014
- [Background] Mazmanian SK, Round JL, Kasper DL. A microbial symbiosis factor prevents intestinal inflammatory disease. Nature. 2008 May 29;453(7195):620-5. doi: 10.1038/nature07008. PMID 18509436
- [Background] Minemura M, Shimizu Y. Gut microbiota and liver diseases. World J Gastroenterol. 2015 Feb 14;21(6):1691-702. doi: 10.3748/wjg.v21.i6.1691. PMID 25684933
- [Background] Roderburg C, Luedde T. The role of the gut microbiome in the development and progression of liver cirrhosis and hepatocellular carcinoma. Gut Microbes. 2014 Jul 1;5(4):441-5. doi: 10.4161/gmic.29599. Epub 2014 Jul 9. PMID 25006881
- [Background] Schnabl B. Linking intestinal homeostasis and liver disease. Curr Opin Gastroenterol. 2013 May;29(3):264-70. doi: 10.1097/MOG.0b013e32835ff948. PMID 23493073
- [Result] Galina V. Fedotovskikh, Galija M. Shaymardanova, Manarbek B. Askarov, Maiya S.Zhumabaeva, Gulmira S. Dosataeva, Aigerim K. Smagulova, Sapargul Marat, Tatyana G. Ezhelenko. Efficiency of mesenchymal stem cell therapy in ulcerative colitis as assessed by the morphology of colon mucosa. J.Cellular Therapy and Transplantation.Vol.8,№2,2019,58-62.